CLINICAL TRIAL: NCT06112288
Title: The Acute Effect Comparisons of Manual Therapy Application to Ankle Soft Tissues or To Ankle Joint on Ankle Motion, Functional Status, and Passive Mechanical Properties of Muscle in Individuals Who Had Achilles Tendon Repair
Brief Title: The Acute Effect Comparisons of Manual Therapy Or Ankle Motion in Individuals Who Had Achilles Tendon Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fırat Tan, Director, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Achilles2023
Record Dates: First submitted 2023-09-29; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Achilles Tendon Rupture; Functional Performance

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive myofascial release (cmr) (Experimental): Participants in the CMR group were instructed to lie prone on the treatment table with their feet off the end of the table. The clinician began the treatment by bending the knee to 90° and shaking the muscle belly of the triceps surae group for 30 seconds. Next, the knee was fully extended, and CMR was performed on the medial and lateral sides of the Achilles tendon for 1 minute, followed by the musculotendinous junction for 2 minutes. Treatment consisted of broad strokes applied with the clinician's knuckles to release superficial restrictions, followed by more specific strokes applied with the clinician's thumb to any located restrictions. Strokes were applied at a contact point of 45° to the tissue, with pressure directed from distal to proximal. At the end of the intervention, the clinician shook the belly of the triceps surae complex for 30 seconds. The same examiner (T.S.) applied all CMR treatments.
  Interventions: Other: Compressive Myofascial Release
- ankle mobilization (Experimental): The joint mobilization group received two sets of ankle joint mobilizations. Each set consisted of two-minutes of Grade III anterior-to-posterior talocrural joint mobilizations with a one-minute rest between sets with the patient in a long-sitting position. This mobilization was operationally defined as large-amplitude, one-second rhythmic oscillations from the mid- to end ROM with translation taken to tissue resistance
  Interventions: Other: Ankle mobilisation

INTERVENTIONS:
Other: Compressive Myofascial Release — Compressive myofascial release is manual therapy technics.
  Arms: Compressive myofascial release (cmr)
Other: Ankle mobilisation — ankle mobilization is manual therapy technics.
  Arms: ankle mobilization

SUMMARY:
Achilles tendon rupture is common among physically active individuals. Limitations, decreases in the level of standing on heel rise, and due to these limitations, failures in functional activities such as returning to sports, walking, running, jumping and performance tests are observed. Manual therapy methods included in rehabilitation programs are an effective option in solving these problems. The aim of the study is to investigate the effects of Compressive Myofascial Release and Ankle joint mobilization on ankle joint movement, functional tests, elasticity and stiffness of the muscle-tendon complex and muscle tone parameters in individuals who underwent Achilles tendon repair.

DETAILED DESCRIPTION:
Achilles tendon rupture is common among physically active individuals. It has been reported that 73% of all Achilles tendon ruptures are sports-related and injuries frequently occur between the ages of 30-49. Conservative or surgical treatments can be applied after Achilles tendon ruptures. After Achilles tendon injuries and repair, decreases in Soleus muscle strength and endurance, changes in lower extremity muscle activation levels, decreases in Gastro-Soleus muscle circumference, increase in Achilles tendon thickness and stiffness, decreases in elasticity, elongations in the Achilles tendon, ankle dorsiflexion range of motion. Limitations, decreases in the level of standing on heel rise, and due to these limitations, failures in functional activities such as returning to sports, walking, running, jumping and performance tests are observed. Manual therapy methods included in rehabilitation programs are an effective option in solving these problems. The aim of the study is to investigate the effects of Compressive Myofascial Release and Ankle joint mobilization on ankle joint movement, functional tests, elasticity and stiffness of the muscle-tendon complex and muscle tone parameters in individuals who underwent Achilles tendon repair. Compressive myofascial release will be applied to a group that has undergone Achilles tendon repair surgery, and ankle mobilization will be applied to another group. Muscle-tendon passive mechanical properties will be evaluated with Myoton-3 before and after the applications. Toe elevation level, ankle joint range of motion and Achilles tendon rest angle will be evaluated before and after the application.

ELIGIBILITY:
Inclusion Criteria:

* • Being male between the ages of 18-55,

  * Having unilateral Achilles tendon repair performed for at least 6 months,
  * No open wound,
  * No history of fracture accompanying Achilles injury.

Exclusion Criteria:

* • Presence of a history of repeated Achilles tendon rupture,

  * Having a rupture or tendon injury on the contralateral side,
  * Having a neurological deficit,
  * Having a history of injury in any of the lower extremity joints for the last 1 year,
  * Having a history of surgery other than Achilles tendon repair in any of the lower extremities,
  * Having a history of corticosteroids applied to the Achilles tendon,

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Passive Mechanical Properties | 2 year
  The device measures the stiffness value in Newtons/meter (N/m).The MG measurement site was located at 30% of the length between the popliteal fossa and lateral malleolus, where cross-sectional areas of the gastrocnemius are almost maximum. LG stiffness was measured at one-third of the length between the small head of the fibula and the heel (Masood et al., 2014). stiffness measurements were performed when participants were in a prone position with the knee joint fully extended and the hip in the neutral position.The probe of the Myoton3 was placed perpendicular to the surface of the soft tissue for the stiffness measurement.

SECONDARY OUTCOMES:
Achilles tendon resting angle (ATRA) | 2 year
  The ATRA test assesses ankle mobility with a goniometer, using one arm along the fibula shaft and the other on the fifth metatarsal head. In the heel-rise test, subjects stand on one foot on a 15-cm high box, measuring the distance between the heel and the step as they raise it as high as possible. This is averaged over three trials.
Heel rise test | 2 year
  During heel-rise test performance subjects stood on one foot on a 15-cmhigh, flat box . Ameasuring tape determined the distance between the plantar surface of the heel and the top of the step as subjects attempted to raise their heel as high as possible and hold this position for 5 seconds. The bony calcaneal prominence where the central Achilles tendon made insertion was palpated to confirm the tape measure placement point. Three test trials were performed, and the average distance was determined.
WBLT (weight bearing lunge test) | 2 year
  Closed kinetic chain ankle dorsiflexion movement magnitude was measured using the WBLT. During WBLT performance, subjects stood barefoot, facing a wall with the test foot parallel to a tape measure placed on the floor. While in this position the opposite foot was placed approximately 1 foot length behind the test foot while maintaining test foot and knee perpendicular alignment with the wall. Subjects performed an anterior lunge with the goal of lightly touching their patella to the wall while keeping their heel firmly planted on the floor. While in this position, the test foot was progressively moved away from the wall in approximately 1-cm intervals, and the test was repeated. This process continued until heel contact could no longer be maintained. At this point, the distance between the distal big toe and the wall was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Güney Deniz, Proffessor, Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Fırat Tan, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No